CLINICAL TRIAL: NCT06357143
Title: Efficacy of Early Multimodal Physiotherapy in Patients With Reverse Shoulder Prosthesis: a Randomized Controlled Trial.
Brief Title: Efficacy of Early Multimodal Physiotherapy in Patients With Reverse Shoulder Prosthesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REMOVE
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Fractures; Prosthesis User
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL GROUP - STANDARD PHYSIOTHERAPY (Active Comparator): Patients will undergo standard care which consists of an initial consultation with the physiotherapist to receive some recommendations about exercises, progression and health education
  Interventions: Other: CONTROL
- EXPERIMENTAL GROUP - REMOVE PROGRAM (Experimental): INITIAL STAGE:
  * Aim: Recover mobility
  * Exercises: Passive therapy, isometric exercises focused on middle deltoid.
  * Goal: 80º passive flexion, 45º abduction, 5 N of abduction force STRENGTHENING STAGE
  * Aim: Enhance scapulohumeral rhythm and strength rotator cura
  * Exercises: Active-assisted therapy, isotonic exercises between 45-90º of forward flexión and abduction with dumbbells and isometric exercises focused on internal and external rotation.
  * Goal: 100º passive flexion, 90º lateral abduction, 10 N of abduction force INTENSIVE STAGE
  * Aim: Improve motor control and increase cross-sectional muscular área
  * Exercises: Rowe with resistance band, wall push ups, lateral elevation with dumbbles, active external and internal rotation.
  * Goal: 15 N of abduction force FUNCTIONAL STAGE
  * Aim: Develope daily life activities
  * Exercises: Overhead tasks, rowe with Kettlebell, internal and external rotations with resistance bands
  * Goal: 20 N of abduction force
  Interventions: Other: REMOVE

INTERVENTIONS:
Other: REMOVE — INITIAL STAGE:
  * Aim: Recover mobility
  * Exercises: Passive therapy, isometric exercises focused on middle deltoid.
  * Goal: 80º passive flexion, 45º abduction, 5 N of abduction force STRENGTHENING STAGE
  * Aim: Enhance scapulohumeral rhythm and strength rotator cura
  * Exercises: Active-assisted therapy, isotonic exercises between 45-90º of forward flexión and abduction with dumbbells and isometric exercises focused on internal and external rotation.
  * Goal: 100º passive flexion, 90º lateral abduction, 10 N of abduction force INTENSIVE STAGE
  * Aim: Improve motor control and increase cross-sectional muscular área
  * Exercises: Rowe with resistance band, wall push ups, lateral elevation with dumbbles, active external and internal rotation.
  * Goal: 15 N of abduction force FUNCTIONAL STAGE
  * Aim: Develope daily life activities
  * Exercises: Overhead tasks, rowe with Kettlebell, internal and external rotations with resistance bands
  * Goal: 20 N of abduction force
  Arms: EXPERIMENTAL GROUP - REMOVE PROGRAM
Other: CONTROL — Patients will undergo standard care which consists of an initial consultation with the physiotherapist to receive some recommendations about exercises, progression and health education
  Arms: CONTROL GROUP - STANDARD PHYSIOTHERAPY

SUMMARY:
The present study try to evaluate the effectivenness of an early intervention program based on multimodal physiotherapy and focused on therapeutic exercise to improve the results of patients with a reverse shoulder phrostesis. This trial will be a randomized controlled trial with parallel groups, and outcomes variables will include psychometric properties through the use of specific questionnaries, and laboratory variables such as strength with a dynamometer, range of movement with a goniometer, muscle mass with an ultrasound, and kinematic parameters with inertial sensors. This study aims to develop an original intervention program in order to try to establish new protocols in the management of these patients.

DETAILED DESCRIPTION:
Background: Shoulder fractures, shoulder osteoarthritis and rheumatoid arthritis have a high prevalence and many times they require a surgery, in which a reverse shoulder phrostesis is colocated. Nonetheless, nowadays there is no a clear consensus protocol in order to manage the prehabilitation and rehabilitation of this patient, so each physiotherapist use different techniques to treat this pathology.

Objective: This study aims to evaluate the effectiveness of an original intervention program (REMOVE program) focused on an early intervention based on therapeutic exercise, manual therapy and education to improve the functionality of these patients after surgery.

Methods: This study is a randomized controlled trial with parallel groups. The control group receive standard care, and the experimental group is subjected to the REMOVE program. Both groups are evaluated five times, pre-surgery, at baseline, at 6 weeks, at 12 weeks and at 24 weeks to assess psychometric and laboratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a reverse shoulder prosthesis.
* Age between 18 and 90 years.
* Signed informed consent.

Exclusion Criteria:

* Language or cultural barriers.
* Other upper limb injury.
* Treatment that affect physical activity capacity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons Scale (ASES) - Functionality. | BASELINE, 12 WEEKS, 24 WEEKS
  This tool is used to evaluate functionality and shoulder-related problems. This scale contains demographic data, medical evaluation, and self-reported outcomes, with a visual analog scale (VAS) to report pain, and 10 items regarding daily life activities.
  The score is calculated: [(10 - score obtained in VAS) x 5] + (5/3 x score obtained in daily life activities)]. The worst result is 0 points and the best one is 100 points.

SECONDARY OUTCOMES:
Ultrasound image - Muscle thickness in centimeters. | BASELINE, 12 WEEKS, 24 WEEKS
  To measure the thickness of lateral deltoid muscle at rest, at maximum contraction, and fatigued, being able to compare the muscle mass variation between presurgical and postsurgical situation, and the effect of the intervention in this variable.
Inertial sensors - Linear acceleration and angular velocity | BASELINE, 12 WEEKS, 24 WEEKS
  To assess kinematics variables such as angular velocity and linear acceleration during flexion, abduction and scaption, to evaluate the scapulohumeral rhythm and the tridimensional scapula motion.
Dynamometer - Strength in Newtons. | BASELINE, 12 WEEKS, 24 WEEKS
  To measure strength, time to peak, rate of force development, and muscle power of the lateral deltoid.
Goniometer - Range of motion in degrees. | BASELINE, 12 WEEKS, 24 WEEKS
  To measure the range of motion, both passive and active, in flexion, abduction, external rotation and internal rotation.
Constant-Murley Score (CS) - Functionality | BASELINE, 12 WEEKS, 24 WEEKS
  To evaluate functional status of the shoulder. The scale is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion (40 points).
  The total score is between 0 points (worst result) and 100 points (best result).
University of California - Los Angeles Shoulder Scale (UCLA) - Functionality. | BASELINE, 12 WEEKS, 24 WEEKS
  To assess functional outcomes after shoulder interventions. The scale include five categories: active forward flexion (5 points), strength of forward flexion (5 points), pain (10 points), satisfaction (5 points), and function (10 points).
  The total score range from 0 points (worst result) and 35 points (best result).
Simple Shoulder Test (SST) - Functionality. | BASELINE, 12 WEEKS, 24 WEEKS
  To evaluate the ability of the affected shoulder to perform daily live activities.
  The tool is based on 12 "yes" (1 point) or "no" (0 points) questions. Overall score is calculated by: [number of "yes" / number of completex items] x 100, were 0 % is the worst result, and 100% is the best result.
Physiological fatigue - high density electromyography | Baseline, 6 Weeks, 12 weeks, 24 weeks.
  We are going to use a matrix of 64 electrodes located on middle deltoid muscle. The variables extracted will be: impulse train, motor neuron recruitment,, neural drive speed
Kinematics - Motion capture system | Baseline, 6 weeks, 12 weeks, 24 weeks.
  We are going to record analytical movements (forward flexion, lateral abduction, scaption) and functional movements with a mobile phone camera, to analyze position, linear acceleration and angular velocity

IPD SHARING:
Plan to Share IPD: No